CLINICAL TRIAL: NCT04519073
Title: Randomized, Placebo-controlled, Double-blind, Phase 1, Dose-escalating Study to Evaluate the Safety and Immunogenicity of a Synthetic Virus Like Particle (SVLP) Vaccine Against Respiratory Syncytial Virus (RSV)
Brief Title: Phase 1 Study to Evaluate the Safety and Immunogenicity of a Candidate Vaccine Against Respiratory Syncytial Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virometix (Industry)
Collaborators: Center of Vaccinology, Ghent, Belgium (CEVAC) (Unknown); Expert Clinical Services Organization, Brussels, Belgium (ECSOR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: VMXRSV306-001
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Acute Bronchiolitis Due to Respiratory Syncytial Virus

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, sequential, parallel cohorts, dose-escalation (three dosages) study in one centre.
Who Masked: Participant, Investigator
Masking Description: The Investigator, the laboratory and the subjects will be kept blind to the treatment arm (placebo/vaccine) to which the subject has been allocated up to the end of the study (Month 12).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 0.5 mL of diluent (phosphate buffer)
  Interventions: Biological: V-306 candidate vaccine
- V-306 low dose (Experimental): V-306 at 15 µg
  Interventions: Biological: V-306 candidate vaccine
- V-306 intermediate dose (Experimental): V-306 at 50 µg
  Interventions: Biological: V-306 candidate vaccine
- V-306 high dose (Experimental): V-306 at 150 µg
  Interventions: Biological: V-306 candidate vaccine

INTERVENTIONS:
Biological: V-306 candidate vaccine — Each V-306 monomer consists of the following elements:
  1. A Lipopeptide Building Block that contains an optimized, artificially designed coiled-coil domain, which self-assembles into highly stable trimers.
  2. A 'universal' T-helper epitope fused at the C-terminus of the coiled-coil domain.
  3. A lipid component di-palmitoyl-S-glyceryl cysteine (Pam2C), fused at the N-terminus.
  4. A mimetic of the Palivizumab epitope, referred to RSV F-protein site II antigen mimetic (FsIIm), which is coupled near the C-terminus of the Lipopeptide Building Block via a short maleimide-PEG-oxime linker.

SUMMARY:
The primary and secondary objectives of this Phase 1 study are respectively to assess the safety and the immunogenicity of two administrations of the RSV vaccine candidate at three different doses.

The study has a randomized, placebo-controlled, double-blind, sequential, parallel cohorts, dose-escalation (three dosages) design. Each of the three cohorts (N=20 subjects per cohort, total of 60 subjects) will receive placebo (n=5), or a low (15 µg, n=15), intermediate (50 µg, n=15) or high dosage (150 µg, n=15) of candidate vaccine, on two occasions (Day 0 and Day 56). Subjects will be healthy adult women aged between 18 and 45 years.

There will be two phases: an active treatment phase from Day 0 to Month 3, and a follow-up phase from Month 3 + 1 day to Month 12.

During the active phase, subjects will complete diary cards to record oral temperature (daily), solicited local and general adverse events (AEs) and unsolicited AEs for 7 days after each administration. Unsolicited AEs will be recorded up to Day 28 post-each administration. Serious adverse events (SAEs) and adverse events of specific interest (AESI) will be recorded throughout the duration of the active phase. Subjects will visit the clinical site for safety monitoring on Days 1, 7 and 28 following each administration.

Blood will be drawn at a screening visit and the safety test data will be available just before 1st administration. The screening set includes markers of infection with hepatitis B virus, hepatitis C virus and human immunodeficiency virus. A serum sample will be taken for detection of pregnancy. At the next scheduled time points, pregnancy will be screened in a urine sample. Laboratory safety parameters will be examined further at Days 0, 1, 7, 28, 56, 57, 63 and 84.

During the follow-up phase, visits for safety monitoring are scheduled at Months 6, 9 and 12 post-1st administration. SAEs and AESI will be recorded at each visit.

Humoral immunity will be measured on Days 0, 28, 56, Month 3, Month 6, Month 9 and Month 12. Cellular immunity will be measured on Days 0, 7, 28, 56, 63 and 84.

The duration of the study for each subject will be approximately 13 months. The total duration of the study will be approximately 18 months.

DETAILED DESCRIPTION:
Virometix designed and developed a candidate vaccine coded V-306 based on synthetic virus like particles (SVLP) that present the neutralizing Palivizumab epitope of the antigenic site II region of the F-protein (FsII). V-306 has been evaluated in cotton rats, mice and rabbits for safety and immunogenicity. Strong immunogenicity was demonstrated in mice and rabbits by ELISA and RSV A and B neutralization. Full protection with no vaccine-associated enhanced respiratory disease (VAERD) was demonstrated in a validated mouse challenge model. Reduction of the viral load with no VAERD was also shown in the cotton rat challenge model.

The primary objective of the first-in-human Phase 1 study is to assess the safety of two administrations of the RSV vaccine candidate at three different dosages of V-306.

The secondary objective is to assess the immunogenicity of two administrations of the RSV vaccine candidate at three different dosages of V-306.

The study has a randomized, placebo-controlled, double-blind, sequential, parallel cohorts, dose-escalation (three dosages) design. It will be conducted in one centre. Each of the three cohorts (N=20 subjects per cohort, total of 60 subjects) will receive placebo (n=5), or a low (15 µg/administration, n=15), intermediate (50 µg/administration, n=15) or high dosage (150 µg/administration, n=15) of candidate vaccine, on two occasions (Day 0 and Day 56). Subjects will be healthy adult women aged between 18 and 45 years. The enrolment schedule with sentinel dosing will be the same in each cohort. After each administration, the subject will be observed in the clinical trial centre for 120 minutes, before being discharged.

The study will be in two phases: (1) an active treatment phase from Day 0 to Month 3, i.e. one month post 2nd administration, with unblinding and primary analysis of data collected up to Month 3, and (2) a follow-up phase from Month 3 + 1 day to Month 12 post-1st administration for safety and immunogenicity. The sponsor will be unblinded at Month 3, while the clinical site and laboratory will remain blinded during the whole study.

During the active phase, subjects will complete diary cards to record oral temperature (daily), solicited local and general adverse events (AEs) and unsolicited AEs for 7 days after each administration. Unsolicited AEs will be recorded up to Day 28 post-each administration. Serious adverse events (SAEs) and adverse events of specific interest (AESI) will be recorded throughout the duration of the active phase. Subjects will visit the clinical site for safety monitoring on Days 1, 7 and 28 following each administration. A time window will be defined for each visit.

Blood will be drawn at a screening visit (up to 14 days before Day 0 for lab safety analyses and up to 2 months before Day 0 for serology analyses) and the safety test data will be available just before 1st administration. The screening set includes markers of infection with hepatitis B virus, hepatitis C virus and human immunodeficiency virus. These data will be part of the baseline health status of each subject. A serum sample will be taken for detection of pregnancy. At the next scheduled time points, pregnancy will be screened in a urine sample and if positive will be confirmed by blood analysis. Laboratory safety parameters will be examined further at Days 0, 1, 7, 28, 56, 57, 63 and 84.

During the follow-up phase, visits for safety monitoring are scheduled at Months 6, 9 and 12 post-1st administration. SAEs and AESI will be recorded at each visit.

Humoral immunity will be measured on Days 0, 28, 56, Month 3, Month 6, Month 9 and Month 12. Months 6, 9 and 12 aim to evaluate the persistence of the humoral response.

Cellular immunity will be measured on Days 0, 7, 28, 56, 63 and 84. Data collection will use an electronic Case Report Form (eCRF). The duration of the study for each subject will be approximately 13 months. The total duration of the study will be approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Healthy women aged between 18-45 years.
* No evidence of disease based on medical history, physical examination, vital signs (blood pressure, heart rate, body temperature and respiratory rate), laboratory safety parameters and clinical judgement.
* Not pregnant and committed to not becoming pregnant during the whole study period. Committed to use adequate and effective contraception means in accordance with the Clinical Trial Facilitation Group (CTFG) criteria.
* The subjects must have used adequate and effective contraception means (CTFG criteria) for at least 60 days prior to the 1st administration.
* Capability to meet the requirements of the study.

Exclusion Criteria:

* Presence of serologic markers of acute or chronic Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBsAg and anti-HBc) and Hepatitis C Virus (anti-HCV) infection(s).
* As judged by the Investigator, any clinically significant disease related to the cardiovascular (CV), gastrointestinal (GI) or central nervous system (CNS).
* Any chronic disease, or history of significant disease that might interfere with the trial's conduct or completion. Some conditions may be accepted if stabilised, e.g. hypertension.
* An active respiratory disease or symptoms thereof (chronic obstructive pulmonary disease, asthma, asthmatic bronchitis, dyspnoea, wheezing, severe allergy) requiring medication, or history of such disease.
* Personal history of active or past autoimmune disease
* Administration for more than three months prior of study start of immunosuppressant or immuno-modifying drugs (including systemic corticosteroids).
* Confirmed or suspected (at the discretion of the Investigator) immuno-suppressive or immuno-deficient condition.
* Current smokers (more than 10 cigarettes/day).
* Blood transfusion, blood product, immunoglobulins received during the period of 3 months prior to study start.
* Clinically significant (according to Investigator's judgement) laboratory out of range values. The abnormal lab test can be neglected if its cause is evident and of no clinical relevance
* Acute disease and/or fever (≥38°C measured by the oral route) at the time of test article administration. Vaccine administration can be postponed until the febrile episode is over.
* Recent vaccination (e.g., vaccine administration within 2 weeks or 4 weeks [live attenuated]) or evidence that a vaccine will be required during the study period (e.g., planned travel).
* Pregnant or plan to become pregnant during the study period.
* Breastfeeding.
* Women highly exposed to children less than 5 years of age will be excluded to reduce risk of RSV infection, including mothers of young children, paediatric nurses, personnel of day nursery.
* Previous participation in a RSV vaccine study.
* Any other significant finding that would increase, according to the Investigator, the risk of having an adverse outcome from participating in the study.
* History of (suspected) hypersensitivity reaction that could be triggered by any component of the vaccine.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Solicited local and general adverse events | During 7 days post-each administration
  Number and percentage of subjects reporting solicited local and general AEs reported on diary card during 7 days post-each administration in the placebo group and in the three vaccine cohorts. Local solicited symptoms are pain, induration, erythema, and swelling at administration site. General solicited symptoms are headache, fatigue, body temperature (measured orally) and generalized myalgia.
Adverse events of special interest (AESI) | Day 0 to Month 12
  Number and percentage of subjects reporting AESI in the placebo group and in the three vaccine cohorts. Monitoring of AESI will include lower respiratory tract infection (LRTI) and respiratory events such as dyspnoea, wheezing, cough, other asthmatic symptoms and increased sputum production.
Serious adverse events | Day 0 to Month 12
  Number and percentage of subjects reporting serious adverse events in the placebo group and in the three vaccine cohorts.

SECONDARY OUTCOMES:
Humoral immune response | Day 0 to Month 12
  RSV micro-neutralization titers against RSV A and B.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sumeray, MD, Study Director — Virometix
Locations (1):
- Centre for Vaccinology (CEVAC), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No